CLINICAL TRIAL: NCT06286735
Title: Effects of Cinnamomum Supplementation on Inflammation, Oxidative Stress, and Intestinal Microbiota in Patients With CKD.
Brief Title: Effects of Cinnamomum Supplementation in Chronic Kidney Disease Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DeniseMafra18
Record Dates: First submitted 2024-02-11; First posted 2024-02-29 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Diseases
Keywords: cinnamomum; chronic kidney diseases; Inflammation; Oxidative stress; Gut microbiota; Biochemical markers
MeSH Terms: conditions — Renal Insufficiency, Chronic; Inflammation | interventions — camphorin protein, Cinnamomum camphora

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): 60 capsules of 500 mg of powdered cinnamomum bark (cinnamomum verum; 40% polyphenols) each. Participants in this group will be instructed to consume two capsules per day, one after lunch and the other after dinner for 3 months.
  Interventions: Dietary Supplement: cinnamomum
- Placebo (Placebo Comparator): 60 capsules with 500 mg of corn starch each. Participants in this group will be instructed to consume two capsules per day, one after lunch and the other after dinner for 3 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: cinnamomum — 60 capsules of 500 mg of powdered cinnamomum bark (Cinnamomum verum; 40% polyphenols). Participants in this group will be instructed to consume two capsules per day, one after lunch and one after dinner for 3 months.
  Arms: Intervention
Other: Placebo — 60 capsules with 500 mg of corn starch per month, until the end of the three months of intervention. Participants in this group will be instructed to consume two capsules per day, one after lunch and the other after dinner for 3 months.
  Arms: Placebo

SUMMARY:
Patients with chronic kidney disease (CKD) experience many complications related to inflammation and oxidative stress that are closely related to the progression of kidney failure and increased mortality. Furthermore, these patients may have intestinal dysbiosis associated with persistent uremia, generating greater production of uremic toxins arising from the metabolism of intestinal bacteria and also helping to maintain the inflammatory process and oxidative stress. In this context, some nutritional strategies have been proposed as an adjuvant therapeutic alternative to modulate inflammation and improve the antioxidant response of patients with CKD, and even more so to modulate the intestinal microbiota. Based on the consolidated knowledge of the role of nutrients and bioactive compounds on the expression of genes related to inflammation, oxidative stress, and also the modulation of the intestinal microbiota, cinnamon, a member of the Lauraceae family, has been widely used as a spice and traditional herbal medicine for centuries and has indicated beneficial benefits in cardiovascular diseases, obesity, diabetes. The bioactive compounds in cinnamomum, such as cinnamaldehyde, cinnamic acid, and cinnamate, can attenuate oxidative stress, inflammation, hyperglycemia, intestinal dysbiosis, and dyslipidemia, which are common complications in CKD patients. Therefore, the present project proposes a longitudinal clinical trial study that aims to evaluate the effects of cinnamomum on transcription factors and inflammatory markers, oxidative stress and modulation of intestinal health in patients with CKD on hemodialysis.

DETAILED DESCRIPTION:
This is a longitudinal study of the randomized, double-blind, placebo-controlled clinical trial type (randomized controlled trial - RCT) where patients will be allocated into two groups [intervention group (15 patients on conservative treatment and 15 patients on hemodialysis ) and placebo group (15 patients on conservative treatment and 15 patients on hemodialysis)]. In the intervention group, participants will receive a capsule containing 60 capsules of 500 mg of powdered cinnamomum bark (cinnamomum verum; 40% polyphenols). Participants in this group will be instructed to consume two capsules per day, one after lunch and the other after dinner for 3 months, and every month the research team will provide a bottle containing 60 capsules of 500 mg of cinnamomum bark powder. (Cinnamomum verum; 40% polyphenols). The placebo group will receive 60 capsules with 500 mg of cornstarch per month, until the end of the three months of intervention, and the guidelines will be the same as those given to the intervention group.

Randomization will be performed after inclusion and exclusion criteria are verified. Eligible patients will be assigned 1:1 to both study arms according to a computer-generated list of treatment codes. An independent, appropriately trained statistician will assign participants to intervention and placebo groups at random. Randomization and allocation will be concealed from researchers and participants until main analyzes are completed.

Blood tests, assessment of food intake and anthropometric measurements will be carried out at the beginning of the follow-up and at the end of three months of treatment, with no additional need for the patient to travel to the collection sites. This will be carried out on hemodialysis days or pre-scheduled routine appointments. If extra travel is necessary, the patient will be reimbursed for transportation costs. Each month, researchers will go to the hemodialysis clinic to check adherence to treatment by counting capsules and subsequently delivering new pots for use in the following month, until the three months of study are completed. In addition, researchers will contact participants by phone weekly to monitor possible side effects, possible questions, and adherence.

ELIGIBILITY:
Inclusion Criteria:

* patients with CKD undergoing conservative treatment stages G3a-G4
* patient in stage 5 (GFR < 15 mL/min), undergoing hemodialysis for more than 6 months and having an arteriovenous fistula (AVF) as vascular access.

Exclusion Criteria:

* pregnant, lactating, smoker patients
* patients using antibiotics in the last 3 months, antioxidant supplements and habitual cinnamon intake
* patients with autoimmune and infectious diseases, cancer, liver disease and AIDS, illiterate people and people with disabilities (visual, hearing)
* patients who are allergic or intolerant to the components of the capsules.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-22 (Estimated); Primary Completion 2025-11-22 (Estimated); Study Completion 2026-12-22 (Estimated)

PRIMARY OUTCOMES:
Concentration of Nuclear factor kappa B (NF-KB) | 3 months
  Inflammation transcription factor

IPD SHARING:
Plan to Share IPD: No